CLINICAL TRIAL: NCT03444714
Title: Phase I Dose-Escalating Study of RiMO-301 With Radiation in Advanced Tumors
Brief Title: Phase I Study of RiMO-301 With Radiation in Advanced Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coordination Pharmaceuticals, Inc. (Industry)
Collaborators: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RiMO-CL17-001
Record Dates: First submitted 2018-02-14; First posted 2018-02-23 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Advanced Tumors
Keywords: intratumoral
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: 3 + 3 dose escalation study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RiMO-301+Radiotherapy (Experimental): 3 dose levels (5%, 10%, and 15% of the total baseline tumor volume, respectively) will be tested in a 3 + 3 dose escalation study
  Interventions: Drug: RiMO-301

INTERVENTIONS:
Drug: RiMO-301 — Drug: RiMO-301 RiMO-301 will be administered by intratumoral route as slow injection
  Radiotherapy Patients will receive 10 fractions of 3 Gy each over 2 weeks
  Other Names: Radiotherapy

SUMMARY:
This is a prospective, open-label, single arm, non-randomized study of RiMO-301 with radiation in patients with advanced tumors. A single escalation dose of RiMO-301 is intratumorally injected in a 3 + 3 study design to identify the recommended dose and dosing volumes.

Condition or Disease:

Patient with advanced tumor which is clinically accessible for intratumoral injection

Intervention/Treatment:

Drug - RiMO-301

Radiation - Radiotherapy

Phase:

Phase 1

DETAILED DESCRIPTION:
Primary Objectives:

• The primary objective is to determine the maximum tolerated dose (MTD) of RiMO-301 as determined by toxicity observed in patients treated with palliative radiation doses

Secondary Objectives:

* To determine clinical response after RiMO-301 and radiotherapy as assessed by clinical response rate using clinical evaluation, imaging and/or symptom relief
* To characterize adverse events of RiMO-301 in patients with advanced cancers
* To evaluate the pharmacokinetics (PK) of RiMO-301 with radiation

The target population is patients with clinically accessible lesions for intratumoral injection. Up to 3 dose levels (5%, 10%, and 15% of the total baseline tumor volume, respectively) will be tested in a 3 + 3 dose escalation study design. MTD will be defined as the dose associated with a dose limiting toxicity (DLT) in less than or equal to 33% of patients at the dose level tested. Dose limiting toxicity (DLT) is defined as one of the following events occurring from the intratumor injection of RiMO-301 to 30 days after the completion of radiation treatment:

* Grade 4 or greater treatment related hematologic or dermatologic toxicity
* Any Grade 3 or greater treatment related non-hematologic, non-dermatologic toxicity (excluding nausea, vomiting or diarrhea without maximal medical intervention)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced or metastatic cancer not amenable to curative therapy
* Lesion that is amenable to palliative radiotherapy
* Lesion that is technically feasible to irradiation and accessible for direct intratumoral injection
* Target tumor in region not in previously irradiated field
* Patient must have recovered from acute toxic effects (≤ grade 1) of previous cancer treatments prior to enrollment
* Age >18 years
* Has measurable disease, defined as at least 1 tumor that fulfills the criteria for a target lesion
* Females with child bearing age should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to the start of dosing
* Patients must sign a study-specific informed consent form prior to study entry

Exclusion Criteria:

* Patients with a histological diagnosis of lymphomas and/or leukemias
* Patients may not have received chemotherapy, targeted therapies, biologic response modifiers and/or hormonal therapy within the last 14 days
* Ongoing clinically significant infection at or near the incident lesion
* Major surgery over the target area (excluding placement of vascular access) <21 days from beginning of the study drug or minor surgical procedures <7 days
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that would make the patient inappropriate for enrollment in this study
* Has any mental or medical condition that prevents the patient from giving informed consent or participating in the trial
* Pregnant and nursing women
* Patients with a target lesion located in a previously irradiated field

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 45 days
  • To determine the maximum tolerated dose (MTD), which is defined as the dose level at which fewer than 33% of patients experience a dose limiting toxicity (DLT) using a 3+3 strategy

SECONDARY OUTCOMES:
clinical benefit | 45 days
  • To assess clinical benefit by change in tumor size and resolution of symptoms, which will be reported as response rate (%)
adverse effect | 45 days
  • To assess adverse effect as either treatment-related or non-treatment-related as defined by CTCAE
Maximum Plasma Concentration [Cmax] | 45 days
  • To evaluate Maximum Plasma Concentration [Cmax] of RiMO-301 in patients tested
Area Under the Curve [AUC] | 45 days
  To evaluate Area Under the Curve [AUC] of RiMO-301 in patients tested

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No
The data will not be shared due to confidentiality agreements